CLINICAL TRIAL: NCT06549231
Title: Evaluation of Efficacy and Safety of Rituximab and Mycophenolate Mofetil Combination in Patients With Interstitial Lung Disease Related to Systemic Sclerosis: a Multicentre Double-blind Placebo-controlled Randomized Trial.
Brief Title: Evaluation of Efficacy and Safety of Rituximab and Mycophenolate Mofetil Combination in Patients With Interstitial Lung Disease Related to Systemic Sclerosis
Acronym: EVER-ILD 3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DR230333
Record Dates: First submitted 2024-07-15; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-06

CONDITIONS: Interstitial Lung Disease With Systemic Sclerosis
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — one course of IV rituximab consisting of an infusion of 1000 mg rituximab (diluted in 500 mL of saline 0.9 % sodium chloride) will be given at day 1, day 15 and an infusion of 500 mg rituximab (in 500 mL of saline 0.9 % sodium chloride) at week 24;
  Arms: Rituximab
Drug: Placebo — one course of intravenous placebo of rituximab consisting of an infusion of 500 mL of saline (0.9% sodium chloride) infusion will be given at day 1, day 15 and week 24;
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy on lung function after 24 weeks of rituximab + MMF combination comparatively to placebo + MMF combination in patients with SSc-ILD severe at the initial assessment or at high risk of progression.

ELIGIBILITY:
Inclusion criteria

1. Male and female 18 years and older who meet the American College of Rheumatology/EUropean League Against Rheumatism collaborative initiative (ACR/EULAR) classification criteria 2013 for systemic scleroderma.
2. Who are eligible for a treatment with MMF (up to 1500 mg twice daily if tolerated) for the management of SSc-ILD adapted from the French PNDS (revised may 2022) [9]:

   * Severe ILD at the baseline assessment i. with an extensive ILD on HRCT ≥20% according to Goh classification [10] ii. or with forced vital capacity of the predicted value (% FVC) ≤ 70%.
   * or ILD regardless of HRCT extension and at high risk of progression (age > 60 years, male gender, early cutaneous diffuse SSc (≤ 5 years), Afro-American or Afro-Caribbean ethnicity, anti-SCL70/Topoisomerase I autoantibody, or biological inflammation with CRP >= 5 mg/L).
   * or ILD regardless of HRCT extension and with progression criteria in the past 6-24 months before the initial assessment (based on INBUILD study): i. relative decline in the forced vital capacity of the predicted value (% FVC) >=10% ii. or relative decline in FVC of 5-10% associated with a relative decline in DLCO >= 15% iii. or relative decline in FVC of 5-10% associated with worsening of dyspnea or extension of ILD lesion on HRCT iv. or worsening of dyspnea with extension of HRCT opacities
3. Person affiliated to a French social security system or equivalent
4. Written informed consent obtained from participant with a specific check box on the Consent form of the study, understanding the risk for men and women treated with mycophenolate mofetil. And additional written consent on the care and contraception agreement form for women of childbearing potential because of use of mycophenolate
5. Ability for subject to comply with the requirements of the study.

   Exclusion Criteria:
6. Known diagnosis of significant respiratory disorders (asthma, tuberculosis, aspergillosis, cystic fibrosis, idiopathic pulmonary fibrosis, sarcoidosis, smoking-related ILD), severe cardiomyopathy or a known severe heart failure as considered by the investigator
7. Known diagnosis of group 1 precapillary pulmonary hypertension (mean pulmonary artery pressure (mPAP) > 20 mmHg and pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg and pulmonary vascular resistance > 2 UWood and FVC ≥ 70% theoretical) or group 3 severe precapillary pulmonary hypertension (mPAP > 20 mmHg and PAWP ≤ 15 mmHg and pulmonary vascular resistance > 5 UWood, whatever the FVC)
8. Concomitant medical or surgical disease, clinically significant as considered by the investigator, serious or unstable, acute or chronically progressive, or any condition that could affect the safety of the patient, in the opinion of the investigator
9. Patient who cannot walk more than 100 meters
10. Known MMF intolerance
11. Initiation of a new therapy for SSc-ILD or with interruption / modification of therapy dosage within 4 weeks prior to baseline assessment
12. Patient having already received a rituximab or MMF-based treatment line for SSc-ILD
13. Known hypersensitivity to rituximab, to murine proteins, other excipients or sulphonamide antibiotics.
14. Concomitant immunosuppressive treatments: >15 mg/day corticosteroids, azathioprine, cyclophosphamide, methotrexate, cyclosporine, tacrolimus, JAK inhibitors within 4 weeks prior to inclusion
15. Treatment with monoclonal antibodies (such as, but not limited to, etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab, tocilizumab) within 6 months prior to inclusion
16. Patients on a lung transplant list
17. Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure: guardianship or trusteeship). Also, women of child-bearing potential (including female partners of sexually active men treated with mycophenolate) not using two reliable contraceptive methods and men not using a contraceptive method (condom), or women and men having a pregnancy project during the year following randomization
18. Patients at high risk of infectious complications: Human Immunodeficiency Virus (HIV) positive or other known immunodeficiency syndromes, hepatitis B and C (HBV, HCV), COVID (within 3 month) or other known viral infection, infection requiring anti-infective treatment within 4 weeks of inclusion
19. Patients with incomplete anti-SARS-CoV-2 vaccine regimen (according to current recommendations) and in this case, patient who has not receive treatment with anti SARS CoV2 therapeutic antibodies (ex : tixagévimab/cilgavimab).
20. Concomitant participation in other interventional research with an investigational drug or medical device.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Forced vital Capacity in % | At 24 weeks
  The primary outcome is the change in Forced Vital Capacity (FVC) (in % predicted) from baseline to week 24 with measures at baseline, week 12 and week 24.

SECONDARY OUTCOMES:
Forced Vital Capacity in % | From baseline to weeks 48
  Change in % of predicted FVC (% FVC)
Forced Vital Capacity in mL | From baseline to weeks 24 and 48
  Change in FVC (mL)
Rodnan skin score | From baseline to weeks 24 and 48
  Change in modified Rodnan skin score (mRSS). This score assesses the extent of thickening at 17 points on the body, simply by palpating the skin. Thickening is from 0 to 3. 0 equals to normal skin thickness and 3 to severe thickening.
Progression free survival | At 24 and 48 weeks
  First event considered
Overall survival | At 48 weeks
Scleroderma Health Assessment questionnaire | From baseline to weeks 24 and 48
  23 questions divided into four groups related to symptoms of vascular, respiratory, gastrointestinal and musculoskeletal dysfunction
King's Brief Interstitial Lung Disease questionnaire | From baseline to weeks 24 and 48
  15 questions about the impact of the disease on life. All answers are from 1 to 7. There is no maximum and minimum.
Living with pulmonary fibrosis symptom questionnaire | From baseline to weeks 24 and 48
  23 questions to evaluate symptoms of pulmonary fibrosis
Living with pulmonary fibrosis impact questionnaire | From baseline to weeks 24 and 48
  21 questions to determine how pulmonary fibrosis affects quality of life.
Diffusing capacity for carbon monoxide | From baseline to weeks 24 and 48
  Changes in % of predicted diffusing capacity for carbon monoxide
6 minutes walk test | From baseline to weeks 24 and 48
  Changes in the 6 minute walk test
Physical activity | From baseline to week 24
  Change in accelerometer-assessed physical activity based on the number of steps per day
Physical activity | From baseline to week 24
  Change in accelerometer-assessed physical activity based on heart rate
Chest image | From baseline to week 48
  Changes in HRCT chest images will be assessed by two thoracic radiologists expert in ILDs, who will score the extent of ILD and the severity of traction bronchiectasis. The ILD extent score will be estimated to the nearest 10% at three lung zones (delimited by the carina and the lowest inferior pulmonary vein for both lungs) and averaged between these 3 zones. Traction bronchiectasis scores will be scored between 0 and 3 (0=absence; 1=mild dilatation without tortuosity; 2=moderate dilatation, < 6mm diameter, with tortuosity; 3=severe dilatation≥ 6mm) for the same three lung zones and averaged for the whole lungs.
Biological markers | From baseline to week 48
  Changes of biological markers related to B-cell depletion. Change in the number of CD19 lymphocytes in absolute value/liter
Biological markers | From baseline to week 48
  Changes of biological markers related to B-cell depletion. Change in the number of CD19 lymphocytes in percentage of leukocytes
Biological markers | From baseline to week 48
  Changes of biological markers related to B-cell depletion. Change in serum gamma globulin concentration in grams/liter
Biological markers | From baseline to week 48
  Changes of biological markers related to B-cell depletion. Change in serum gamma globulin concentration as a percentage of serum proteins
Advers events | From baseline to week 48
  Analyze of all adverse events, especially serious infectious adverse events, occurring during treatment period
Pharmacokinetic | At Day 1, day 15, week 12, week 24 and week 48
  Pharmacokinetic parameters of rituximab : volume of distribution in liter
Pharmacokinetic | At Day 1, day 15, week 12, week 24 and week 48
  Pharmacokinetic parameters of rituximab : clearance in mili liter per minute
Pharmacokinetic | At Day 1, day 15, week 12, week 24 and week 48
  Pharmacokinetic parameters of rituximab : half life in secondes
Cumulative doses of corticosteroids | At week 24 and week 48